CLINICAL TRIAL: NCT07106450
Title: Muscle-derived Extracellular Vesicles and Their Interactions With Adipocytes in Human Metabolic Dysfunction
Brief Title: Training Induced Muscle-Adipose EV Communication
Acronym: TIMER2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan Wen (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Yuan Wen, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P20GM156679-Prj5; P20GM156679 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
Keywords: muscle; extracellular vesicles; adipose
MeSH Terms: conditions — Prediabetic State | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute Resistance Exercise (Experimental): Participants will perform four exercises: squat, knee extension, leg press, and lat pulldown at 80% of 1-RM (repetition maximum) determined during a previous visit.
  Interventions: Behavioral: Acute Resistance Exercise

INTERVENTIONS:
Behavioral: Acute Resistance Exercise — Participants will perform three sets of eight repetitions, with a 90-120 second rest between sets, with a fourth set performed to failure. All resistance exercise will be performed on pneumatic resistance devices (Keiser Sports Health Equipment, Fresno, CA).
  Other Names: Strength Training

SUMMARY:
This study examines how muscle cells communicate with fat cells through tiny packages called extracellular vesicles (EV) during exercise. These vesicles carry important molecules that may affect how the body processes sugar and fat. The research team observed significant variability in the adipose response to exercise, and used this variability to gain further insight into the mechanism through which mature microRNA-1 (miR-1) changes in adipose tissue. The investigators selected six subjects with the highest increase in miR-1 abundance in adipose tissue after exercise and compared them with the six subjects that had the most dramatic decrease in miR-1 abundance after exercise. The research team observed that participants intrinsically vary in their ability to endocytose EV into adipose tissue. It is unclear whether this variance in receptivity is a cause or consequence of the significant difference in EV-delivery of miR-1 to adipose tissue.

DETAILED DESCRIPTION:
This study investigates muscle-derived extracellular vesicle (EV) communication with adipose tissue and how this pathway is altered in pre-diabetes. The investigators will recruit 80 participants (40 euglycemic controls, 40 pre-diabetic) aged 18-30 years, equally distributed by sex. Pre-diabetes will be defined as impaired fasting glucose (100-125 mg/dL), impaired glucose tolerance (2-hour oral glucose tolerance test (OGTT) 140-199 mg/dL), or HbA1C 5.7-6.4%.

Following informed consent and medical screening at the Center for Clinical and Translational Sciences, participants will undergo baseline blood draw and tissue biopsies (subcutaneous adipose and vastus lateralis muscle) one hour prior to exercise. The resistance exercise protocol consists of whole-body resistance training at 80% 1RM (repetition maximum) intensity including bench press, leg press, and pull-downs. Blood samples will be collected immediately post-exercise and at 30, 60, and 90 minutes. Post-exercise biopsies will be obtained approximately 60 minutes after exercise cessation.

Laboratory analyses will include: (1) microRNA-1 (miR-1) quantification in adipose tissue by quantitative reverse transcription polymerase chain reaction (qRT-PCR) as the primary validated outcome of EV uptake; (2) fluorescently-labeled EV uptake assessment in cultured adipocytes using microscopy; (3) RNA sequencing (RNA-seq) of adipose tissue to identify transcriptomic signatures associated with EV uptake capacity; (4) primary cell culture studies using adult-derived human adipocyte stem cells (ADHASC); and (5) EV isolation and characterization using size exclusion chromatography and density gradient centrifugation.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* Sedentary lifestyle (exercise <1 day/week for at least 3 months prior to enrollment)
* Able to provide informed consent
* For Control Group: BMI < 27 kg/m², normal glucose tolerance, no more than 1 feature of metabolic syndrome
* For Prediabetic Group: BMI > 30 kg/m², at least 3 features of metabolic syndrome including prediabetes (defined as fasting plasma glucose 100-125 mg/dL OR 2-hour post-load glucose on 75g OGTT 140-199 mg/dL OR HbA1C 5.7-6.4%)

Exclusion Criteria:

* Pregnancy (confirmed by pregnancy test in women of childbearing potential)
* Type 2 diabetes mellitus
* Cardiovascular contraindications to resistance exercise
* Medical conditions that would interfere with muscle or adipose tissue biopsy procedures
* Use of medications that significantly affect glucose metabolism or exercise response
* Active participation in structured exercise programs (>1 day/week) within 3 months of enrollment
* Inability to safely participate in resistance exercise protocol

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
miR-1 abundance in adipose tissue | 60 minutes post-exercise (single measurement)
  Quantification of mature microRNA-1 levels in subcutaneous adipose tissue biopsies using quantitative Real Time-PCR as validated biomarker of in vivo extracellular vesicle uptake
Extracellular vesicle uptake capacity in primary adipocytes | 24-48 hours post-isolation (in vitro culture)
  Measurement of fluorescently-labeled extracellular vesicle internalization in cultured primary adipocytes using confocal microscopy to quantify uptake rates in units of vesicles per minute per cell.

SECONDARY OUTCOMES:
Serum extracellular vesicle miR-1 content | Baseline, 0, 30, 60, and 90 minutes post-exercise
  Time-course analysis of microRNA-1 abundance in isolated serum extracellular vesicles using quantitative RT-PCR to track temporal dynamics of muscle-derived vesicle release
Adipose tissue transcriptomic signatures | 60 minutes post-exercise (single measurement)
  RNA-sequencing analysis of subcutaneous adipose tissue to identify differential gene expression patterns associated with high versus low extracellular vesicle uptake capacity, focusing on endocytotic pathways
Adrenergic receptor gene expression in adipose tissue | 60 minutes post-exercise (single measurement)
  Quantitative RT-PCR measurement of ADRβ1, ADRβ2, and ADRβ3 receptor mRNA levels in subcutaneous adipose tissue as downstream targets of miR-1 delivery
Primary muscle miR-1 transcript levels | 60 minutes post-exercise (single measurement)
  Quantification of pri-miR-1a and pri-miR-1b primary transcript abundance in vastus lateralis muscle biopsies using quantitative RT-PCR to assess exercise-induced miR-1 biogenesis

OTHER OUTCOMES:
Extracellular vesicle tetraspanin marker profiles using ExoView platform | Baseline and 90 minutes post-exercise
  Characterization of circulating extracellular vesicle subpopulations based on surface tetraspanin protein expression (CD63, CD81, CD9) using ExoView R100 platform immunofluorescence detection and high resolution imaging.
  Units of Measure: Percentage of total vesicles positive for each marker.
Circulating extracellular vesicle count using ExoView single vesicle analysis platform | Baseline and 90 minutes post-exercise
  Total number of circulating extracellular vesicles quantified using the ExoView R100 platform single vesicle analysis technology with tetraspanin capture antibodies (CD63, CD81, CD9). Units of Measure: Particles per milliliter
Extracellular vesicle size distribution using ExoView single vesicle analysis | Baseline and 90 minutes post-exercise
  Size characterization of individual circulating extracellular vesicles measured using ExoView R100 platform automated analysis. Units of Measure: Nanometers (diameter).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wen, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality. Summary results and findings will be made available through peer-reviewed publications and presentation at scientific conferences.